CLINICAL TRIAL: NCT02803528
Title: A Comparative Study of the Performance of Biodentine and Mineral Trioxide Aggregate (MTA) in Direct Pulp Capping of Deeply Carious Teeth.
Brief Title: Comparative Study Between Biodentine and Mineral Trioxide Aggregate in Direct Pulp Capping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-OperDent-01-2016
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Patients With Deep Carious Lesions
MeSH Terms: interventions — tricalcium silicate; Pemetrexed

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biodentine (Experimental): The exposed area of the pulp is going to be covered with Biodentine.
  Interventions: Drug: Biodentine
- MTA (Active Comparator): The exposed area of the pulp is going to be covered with MTA
  Interventions: Drug: MTA

INTERVENTIONS:
Drug: Biodentine — Biodentine is going to be used as the direct pulp capping material
  Arms: Biodentine
Drug: MTA — MTA is going to be used as the direct pulp capping material in the second group
  Arms: MTA

SUMMARY:
Comparative study between Biodentine and MTA in direct pulp capping of deeply carious teeth.

ELIGIBILITY:
Inclusion Criteria:

1. asymptomatic vital molars (upper or lower)
2. with complete formation of roots
3. Aged 15 to 30 years.
4. Accidental point pulp exposure during the process of removing dental caries.

Exclusion Criteria:

1. If the molar not vital.
2. If the molar is symptomatic.
3. Immature molar.
4. Patient not in age between (15-30 years).

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
Success at 3 months following capping | the success of treatment is assessed at three months following the application of the material
  Case is considered successful if clinical and radiographic examinations of tooth are sound 100%.
Success at 6 months following capping | the success of treatment is assessed at six months following the application of the material
  Case is considered successful if clinical and radiographic examinations of tooth are sound 100%.
Success at 9 months following capping | the success of treatment is assessed at 9 months following the application of the material
  Case is considered successful if clinical and radiographic examinations of tooth are sound 100%.
Success at 12 months following capping | the success of treatment is assessed at 12 months following the application of the material
  Case is considered successful if clinical and radiographic examinations of tooth are sound 100%.
Success at 18 months following capping | the success of treatment is assessed at 18 months following the application of the material
  Case is considered successful if clinical and radiographic examinations of tooth are sound 100%.
Success at 24 months following capping | the success of treatment is assessed at 24 months following the application of the material
  Case is considered successful if clinical and radiographic examinations of tooth are sound 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad MN Aldakak, DDS MSc, Principal Investigator — PhD Student in Operative Dentistry; Souad Abboud, DDS MSc PhD, Study Chair — Associate Professor of Operative Dentistry, University of Damascus Dental School, Damascus, Syria
Locations (1):
- Department of Operative Dentistry, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guneser MB, Akbulut MB, Eldeniz AU. Effect of various endodontic irrigants on the push-out bond strength of biodentine and conventional root perforation repair materials. J Endod. 2013 Mar;39(3):380-4. doi: 10.1016/j.joen.2012.11.033. Epub 2013 Jan 16. PMID 23402511
- [Background] Iwamoto CE, Adachi E, Pameijer CH, Barnes D, Romberg EE, Jefferies S. Clinical and histological evaluation of white ProRoot MTA in direct pulp capping. Am J Dent. 2006 Apr;19(2):85-90. PMID 16764130
- [Background] Koubi G, Colon P, Franquin JC, Hartmann A, Richard G, Faure MO, Lambert G. Clinical evaluation of the performance and safety of a new dentine substitute, Biodentine, in the restoration of posterior teeth - a prospective study. Clin Oral Investig. 2013 Jan;17(1):243-9. doi: 10.1007/s00784-012-0701-9. Epub 2012 Mar 14. PMID 22411260
- [Background] Laurent P, Camps J, De Meo M, Dejou J, About I. Induction of specific cell responses to a Ca(3)SiO(5)-based posterior restorative material. Dent Mater. 2008 Nov;24(11):1486-94. doi: 10.1016/j.dental.2008.02.020. Epub 2008 Apr 29. PMID 18448160
- [Background] Zanini M, Sautier JM, Berdal A, Simon S. Biodentine induces immortalized murine pulp cell differentiation into odontoblast-like cells and stimulates biomineralization. J Endod. 2012 Sep;38(9):1220-6. doi: 10.1016/j.joen.2012.04.018. Epub 2012 Jul 24. PMID 22892739